CLINICAL TRIAL: NCT00514657
Title: Trial in Periodontal Tissue Regeneration Using Fibroblast Growth Factor-2 (Randomised Controlled Phase II Clinical Trial)
Brief Title: Trial in Periodontal Tissue Regeneration Using Fibroblast Growth Factor-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaken Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KCB-1D-01
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — trafermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- P (Placebo Comparator)
  Interventions: Drug: Trafermin (genetical recombinant of human basic Fibroblast Growth Factor)
- L (Experimental): low dose (0.03 %)
  Interventions: Drug: Trafermin (genetical recombinant of human basic Fibroblast Growth Factor)
- M (Experimental): medium dose (0.1 %)
  Interventions: Drug: Trafermin (genetical recombinant of human basic Fibroblast Growth Factor)
- H (Experimental): high dose (0.3 %)
  Interventions: Drug: Trafermin (genetical recombinant of human basic Fibroblast Growth Factor)

INTERVENTIONS:
Drug: Trafermin (genetical recombinant of human basic Fibroblast Growth Factor)

SUMMARY:
The present clinical trial clarified that basic fibroblast growth factor-2 (FGF-2) can induce regeneration of periodontal tissue lost by progression of periodontitis and evaluated the safety of such induction.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as 2- or 3-walled vertical intrabony defect >=3 mm deep from the top of the remaining alveolar bone
* with mobility of the tooth of degree 2 or less
* with width of attached gingiva appropriate for Guided Tissue Regeneration

Exclusion Criteria:

* concomitant administration of adrenal cortical steroid within 4 wks after the surgery
* administeration of calcium antagonist during the 4 weeks preceding administration of the investigational drug
* coexisting malignant tumour or history of the same
* coexisting diabetes (HbA1C >= 6.5%)
* an extremely poor nutritional condition (serum albumin concentration <2 g/dL)
* pregnancy or lactation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2001-12; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
rate of increase in alveolar bone height | 36 weeks after administration
clinical attachment level (CAL) regained | 36 weeks after administration

SECONDARY OUTCOMES:
time course of rate of increase in alveolar bone height | within 36 weeks after administration
time course of CAL regained | within 36 weeks after administration
the other periodontal inspections (PD, BOP, GI etc.) | within 36 weeks after administration

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Tamura, Ph.D, Study Director — Kaken Pharmaceutical Co., Ltd.

REFERENCES:
- [Derived] Kitamura M, Nakashima K, Kowashi Y, Fujii T, Shimauchi H, Sasano T, Furuuchi T, Fukuda M, Noguchi T, Shibutani T, Iwayama Y, Takashiba S, Kurihara H, Ninomiya M, Kido J, Nagata T, Hamachi T, Maeda K, Hara Y, Izumi Y, Hirofuji T, Imai E, Omae M, Watanuki M, Murakami S. Periodontal tissue regeneration using fibroblast growth factor-2: randomized controlled phase II clinical trial. PLoS One. 2008 Jul 2;3(7):e2611. doi: 10.1371/journal.pone.0002611. PMID 18596969